CLINICAL TRIAL: NCT06211543
Title: Letermovir (LMV) Prophylaxis in CMV-seronegative Allogeneic Stem Cell Transplant Recipients With CMV Seropositive Donors: an Exploratory Study From Spanish GETH/TC Centers
Status: Not yet recruiting | Type: Observational
Sponsor: Grupo Espanol de trasplantes hematopoyeticos y terapia celular (Other)
Responsible Party: Sponsor
Other Study IDs: GETH-LMV
Record Dates: First submitted 2024-01-09; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: CMV
Keywords: CMV; Allogeneic Stem Cell Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LMV cohort: Patients will receive oral or intravenous (if available ) LMV at a dose of 480mg/day. For patients receiving concomitant cyclosporine treatment, the LMV dose will be 240mg/day. LMV will be administered daily through week 14 after transplantation for up to 8 weeks (~Day 100) beginning
- Historical cohort: An historical control cohort for comparison purposes will be used. Historical data will be obtained from a national CMV data base (GETH-GRUCINI), that includes stem cell transplant recipients from September 2014 to December 2022

SUMMARY:
This is an observational cohort study. Two cohort will be enrolled:

LMV cohort: All patients included in in this study will receive LMV according to standard of care.

Historical cohort: an historical cohort will be included to compare the results of both groups (LMV vs historical cohort).

DETAILED DESCRIPTION:
All patients will receive treatment wtith LMV according to standard of care.

Eligible patients will be enrolled in the study under the supervision of the investigator or designated sub-investigators. If possible, patients will receive treatment on an outpatient basis except for the hospitalization requirement established in the protocol.

Patients will receive oral or intravenous LMV (if available) at a dose of 480 mg/day. For patients receiving concomitant treatment with cyclosporine, the dose of LMV will be 240 mg/day. According to the standard of care, LMV will be administered daily until week 14 post-transplant for up to 8 weeks (~day 100) starting on day +1.

Patients could be discontinued earlier if, disease progression, patient withdrawal, loss to follow-up, end of study, or death.

After completion of the treatment period, an end-of-treatment visit will occur within 30 days of receipt of the last dose of study drug.

To compare the outcome of the LMV group, a historical cohort will be selected from the national CMV database (GETH-GRUCINI).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* First allogenic HCT
* Pre-HCT patient CMV negative IgG serology with CMV IgG positive donor serostatus
* Able to provide written consent and complete the informed consent
* Absence of CMV DNAemia requiring antiviral therapy within 5 days before initiation of LMV. Low levels CMVDNAemia before the inception of letermovir are allowed

Exclusion Criteria

* Active pre-emptive therapy for csCMV-I.
* Patients who have received LMV prophylaxis prior to enrollment
* Patients enrolled in a CMV pre-emptive therapy clinical trial
* Glomerular filtration rate (GFR) </=30 mL/min/1.73m^2 (equivalent to creatinine clearance </=10 mL/min)
* Severe hepatic function grade 3-4 CTAE at the time of study entry.
* Suspected or known hypersensitivity to active or inactive ingredients of LMV formulations
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to letermovir.
* Pregnancy or breastfeeding
* Plans to conceive or father children within the projected duration of the trial
* History of current evidence of any condition, therapy, lab abnormality, or other circumstance that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or would place the subject at undue risk as judged by the investigator, such that it is not in the best interest of the subject to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CMV-seronegative Allogeneic Stem Cell Transplant Recipients with CMV seropositive donors
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
CMV DNAemia requiring preemptive treatment or CMV disease | Week 14 post-SCT
  To determinate the incidence of csCMV infection through week 14 post-SCT.

SECONDARY OUTCOMES:
Neutrophile (>0,5x10e9/L) and platelets engraftment (>20 x10e9/L) by day +40 post-SCT. | Day +40 post-SCT
  Engraftment incidence and time to engraftment
Neutrophile (>0,5x10e9/L) and platelets engraftment (>20 x10e9/L) by day +100 post-SCT. | Day +100 post-SCT
  Engraftment incidence and time to engraftment
Death by any cause and death not related with disease relapse or progression | Week 14 post-SCT
  All-cause mortality week 14
Death by any cause non related to relapse | Week 14 post-SCT
  Non-relapse Mortality (NRM)
Death by any cause non related to relapse | Week 24 post-SCT
  Non-relapse Mortality (NRM)
Time to onset of all-cause failure of prophylaxis against CMV infection during the 8 weeks of study-drug administration period (day +100 post-transplant) | Up to 8 weeks of study-drug administration period (day +100 post-transplant)
  To evaluate the time to onset of all-cause failure of prophylaxis against CMV infection during the 8 weeks of study-drug administration period (day +100 post-transplant)
Duration of any CMV-antiviral treatment by day 180 post-SCT | day 180 post-SCT
  To estimate the duration of CMV-antiviral treatments by day 180 post-SCT.
Incidence of blips, clinical and analytic characteristics. | 180 days post-SCT
  To investigate the natural history of blips in the LMV primary prophylaxis (PP) clinical setting
Incidence of untreated CMV DNAemia | 180 days post-SCT
  Incidence of low levels of CMV DNAemia not requiring PET
Adverse events according to the CTCAE, physical examination and regular laboratory tests | 180 days post-SCT
  To evaluate LMV tolerance and safety
Incidence of aGVHD within 120 days after HCT and its onset and severity | 120 days post-SCT
  To evalute de incidence of aGVHD and clinical characteristics.
Incidence of relapse within 180 days after HCT and its onset and severity | 180 days post-SCT
  To evalute de incidence of relapse and clinical characteristics.
Incidence of CMV DNAemia requiring PET within 100-180 days after HCT | From day 100 to day 180 after HCT
  To establish incidence of late (> d +100) clinically significant CMV DNAemia
Incidence of non-CMV infections within 180 days after HCT and its onset and severity | 180 days post-SCT
  To establish de incidence of non-CMV infections.